CLINICAL TRIAL: NCT00637871
Title: Randomised, Double-blind, Placebo Controlled, Parallel-group, Multicentre Phase II Study to Assess Dose Response Relationship of Nolvadex (Oral Tablet) in Prophylactic Treatment of Gynaecomastia and Breast Pain Associated With CASODEX 150 mg (Oral Tablet), and to Assess the Tumour Control…..
Brief Title: Casodex - Nolvadex Combination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7054IL/0044; D6876C00044
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Gynaecomastia; Prostate Cancer
Keywords: Casodex; bicalutamide; Tamoxifen; Gynaecomastia; Prostate Cancer
MeSH Terms: conditions — Gynecomastia; Prostatic Neoplasms | interventions — bicalutamide; Tamoxifen

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Casodex
- 2 (Active Comparator)
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Casodex — 150mg once daily
  Arms: 1
Drug: Tamoxifen
  Other Names: Nolvadex
  Arms: 2

SUMMARY:
This study looks at the relationship in the dose of nolvadex and the incidence of gynaecomastia and also Prostate Specific Antigen (PSA) inhibition when co-administered with Casodex. The aim of the study is to assess the optimal dose of nolvadex which will reduce the breast tissue adverse effects without reducing the efficacy of Casodex.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with adenocarcinoma of the prostate gland but with no evidence of distant metastasis. The stage of disease should be T1-T4, any N, M0 confirmed histologically or cytologically
* Subjects in need of immediate hormonal therapy.
* PSA equal or above 4 ng/ml

Exclusion Criteria:

* Presence of gynaecomastia and/or breast pain at screening visit
* Any previous endocrine therapy for prostate cancer other than neoadjuvant LHRH therapy prior to primary therapy of curative intent.
* Current use, or within the previous 6 months, of any medication known to have a high risk of causing gynaecomastia .
* Previous mastectomy or radiation to chest wall

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

SECONDARY OUTCOMES:
To describe the extent of gynaecomastia and breast pain by treatment group
To describe the relative change from baseline in sex hormones concentrations by treatment group
To describe the pharmacokinetics of tamoxifen, N-desmethyltamoxifen and R-bicalutamide when nolvadex is co-administered at varying doses with CASODEX 150 mg once daily
To assess the tolerance of nolvadex when co-administered at varying doses with CASODEX 150 mg once daily

CONTACTS AND LOCATIONS:
Overall Officials: Yves Fradet, M.D., Principal Investigator — Quebec City